CLINICAL TRIAL: NCT03979170
Title: Patient-derived Organoids of Lung Cancer to Test Drug Response
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Frederic TRIPONEZ, Professor, University Hospital, Geneva
Other Study IDs: 2018-02395
Record Dates: First submitted 2019-04-15; First posted 2019-06-07 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer; Organoid
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Biospecimen retention: blood; cells; tumour tissue for immunohistochemical analysis.
  Tissue of lung cancer will be collected during surgery in a way that will not interfere with subsequent pathological analysis and staging. Under the premise of ensuring normal detection requirements, a certain volume of fresh tumour tissues will be subjected to ex vivo 3-D culture to establish patient-derived tumour organoid models. The lung patient-derived organoids will be characterized. The organs successfully cultured will be kept in liquid nitrogen for at least 10 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Lung tumor resection — lung tumor resection

SUMMARY:
This is a single center, single arm, open and exploratory clinical study, with 50 cases planned for a period of 3 years. The purpose of this study is to evaluate the consistency and accuracy of a Patient-Derived Organoid (PDO) Model of lung cancer to predict the clinical efficacy of anti-cancer drugs, in order to predict the best chemotherapy regimen for each given patient.

DETAILED DESCRIPTION:
The aim of the project is to use a combination of patient-derived organoid models:

* To amplify tumour tissue to obtain enough material for genomic and histological analysis
* to characterize the lung cancer sub-type
* To predict treatment (non)response.

The following points will be addressed:

1. First, the investigators plan to establish and characterize formation of organoids from biopsies of patients with lung cancer: in spheroids, in the 3D cellular model OncoCilAirTM (OncoTheis), and on the chick chorioallantoic membrane (CAM). Patient-derived organoids from tumoural tissue (PDO) will be characterized and compared to the original tumour.
2. Second, the investigators will test the chemoresponse (chemosensitivity and chemoresistance) of organoids to anti-cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven lung cancer
* Age ≥ 18
* Written informed and signed consent
* Accessible to biopsy and/or surgery sample of metastasis and/or primitive tumour

Exclusion Criteria:

* Less than 18 years of age
* Not able to give informed consent (language, intellectual capacities, etc.)
* Not accessible to biopsy and/or surgery sample
* Not enough lung tissue for a histological analysis or the remaining lung tissue is not enough to perform a routine pathological analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients (estimated 50 patients) with histologically proven lung cancer undergoing surgery related to this cancer at the University Hospitals of Geneva.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Patient-derived organoid establishment | 3 years
  Successful generation of lung cancer organoids (growth of lung tumoral cells). The rate of successful generation of lung cancer organoids could vary with the age of the patient, the histological and molecular subtype of lung cancer
Patient-derived organoid validation | 5 years
  Proportion of patient-derived organoids that are histologically and genetically identical to the source tumour

SECONDARY OUTCOMES:
Drug sensitivity | 2019 - 2023
  Drug sensitivity of patient-derived tumour organoids (drug screening and chemotherapy resistance test) Secondary drug effects on patient-derived normal lung organoids
Prediction of the response to treatment by the patient-derived organoids | 2020 - 2025
  The drug sensitivity was tested on patient-derived tumour organoids, which is compared with clinical response of the chemo- or targeted therapy treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mueggler A, Pilotto E, Perriraz-Mayer N, Jiang S, Addeo A, Bedat B, Karenovics W, Triponez F, Serre-Beinier V. An Optimized Method to Culture Human Primary Lung Tumor Cell Spheroids. Cancers (Basel). 2023 Nov 25;15(23):5576. doi: 10.3390/cancers15235576. PMID 38067281